CLINICAL TRIAL: NCT06351189
Title: Performance Evaluation of the NETTI Wheelchair in Dynamic Mode for Subjects With Involuntary Movements With an Impact on Sitting Position Compared With Its Static Mode. Single-case Experimental Design.
Brief Title: NETTI Wheelchair: Does Dynamic Mode or Static Mode Affect the Sitting Position in Patients With Involuntary Movements ?
Acronym: DYNAMIC SYSTEM
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: CIVI/2022/AD-01
Record Dates: First submitted 2024-04-02; First posted 2024-04-08 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-12

CONDITIONS: Hyperextension Spasms; Involuntary Movements
Keywords: Wheelchair; Single-case experimental design; Hyperextension spasms; Positioning
MeSH Terms: conditions — Dyskinesias | interventions — Observation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Control group: STATIC MODE: The patient will be positioned on the Netti Dynamic chair in static mode.
  Interventions: Device: Observation
- Interventional group: DYNAMIC MODE: The patient will be positioned on the Netti Dynamic chair in dynamic mode.
  Interventions: Device: Observation

INTERVENTIONS:
Device: Observation — Patients will be filmed in sitting position in the NETTI DYNAMIC chair, either in static mode or dynamic mode for a period of 3 hours each time.

SUMMARY:
This study compares two modes of the NETTI wheelchair (dynamic or sitting) for patients with hyperkinetic syndromes, to discover which mode is the most comfortable and best suited to these patients.

It is a prospective, single-center pilot study comparing two medical devices evaluated using SCED (Single Case Experimental Design) ABAB methodology: NETTI DYNAMIC chair in dynamic mode (intervention group; phase B) versus the same chair in static mode (control group; phase A). The subject will be his/her own control

DETAILED DESCRIPTION:
Hyperkinetic syndromes are characterized by excessive or involuntary movements throughout the day. These abnormal movements interfere with maintaining the ideal sitting position and cause positioning disorders that may have functional repercussions. To facilitate staying in the ideal position, therapists adapt sitting positions. Together with the patient, they choose the position that appears to be the most functional and comfortable. To maintain this position, the solutions proposed are mainly based on restraint (shells, abduction blocks, straps, etc.). These can be poorly tolerated by the patient, causing discomfort or even pain which can hinder participation. Repeated stresses on the supports, and on the chair itself, leads to frequent breakage. Also, depending on the underlying neurological mechanisms behind the abnormal movements, the question arises as to whether restraint increases the frequency or amplitude of abnormal movements by generating oppositional constraints, areas of discomfort and/or pain, or by reducing functional capacities and frustration caused by these abnormal movements (Cimolin et al. 2009). All these issues can have a significant impact on the quality of life of this population of patients suffering from abnormal movements and who are almost exclusively in wheelchairs. To address these issues, dynamic wheelchair systems have been have been developed to absorb the mechanical stresses generated by abnormal movements.

The chair's dynamic components absorb the force. When the patient's force ceases, the stored energy is returned by the dynamic component which, in turn, helps the patient return to his or her starting position. The ideal seating system enables controlled movement whilst providing mechanical stability.

This is a prospective, single-center pilot study comparing the two medical device modes using an ABAB-type Single Case Experimental Design methodology: The NETTI DYNAMIC chair in dynamic mode (interventional group; phase B) versus the same chair in static mode (control group; phase A). The subject will be his/her own control.

Phase B (intervention) will be performed by positioning the subject on the Netti Dynamic chair in its dynamic configuration. Phase A (control), on the other hand, will be performed positioned on the same chair, but in static mode (backrest and seat locked by means of a jack and pin, legrest and headrest replaced by standard elements and headrest replaced by standard components, making it impossible to adapt the chair's of the chair). In this way, the specific effect of the dynamic mode will be able to be controlled.

The ABAB study design was chosen for this study because it provides the highest level of evidence evidence (Level 1; OCEBM Levels of Evidence Working Group. (2011). "The Oxford 2011 Levels of Evidence." Oxford Centre for Evidence-Based Medicine). It is characterized by the presence of two phases (phase A: control phase and phase B: intervention phase) which are alternated twice.

Each phase must comprise three to five measures to enable reliable statistical analysis. This approach is particularly appropriate for evaluating medical devices, especially when the when the population concerned is heterogeneous. Indeed, an intensive, prospective study of a few individuals, using a methodology defined a priori, including systematic observations, repeated measurements and appropriate data analysis is the most appropriate in this case.

ELIGIBILITY:
Inclusion Criteria:

* Patient with involuntary extension movements with a frequency greater than (>) 3/hour and requiring at least one wheelchair repositioning every 2 hours.
* Patient using a wheelchair and requiring to be in a seated position at least 4 hours per day.
* Patient and/or representative with free and informed consent.
* Patient and/or representative having signed the consent form.
* Patient affiliated or beneficiary of a health insurance plan.
* Patient over 16 years of age (≥16 years).

Exclusion Criteria:

* Patient unable to sit in chair for at least 3 hours a day.
* Patient unable to sit in the chair without the use of a thermoformed corset.
* Patients weighing over 135kg.
* Patient participating in a drug study.
* Patient in an exclusion period determined by another study.
* Patient/legal representative for whom it is impossible to provide informed information.
* Pregnant or breast-feeding patient

Min Age: 16 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: The study population is made up of patients with involuntary extension movements at a frequency of more than 3/hour, requiring at least one wheelchair repositioning every 2 hours, cared for in a medico-educational institute, a specialized residence such as a Specialised Care Home or a Medicalized Care Home, or living at home if necessary.
Sampling Method: Non-Probability Sample
Enrollment: 4 (Actual)
Dates: Start 2024-03-19 (Actual); Primary Completion 2024-12-05 (Actual); Study Completion 2024-12-05 (Actual)

PRIMARY OUTCOMES:
Forward slippage in static mode (PHASE A) | End of the 3-hour period on Day 7
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in static mode (PHASE A) | End of the 3-hour period on Day 14
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in static mode (PHASE A) | End of the 3-hour period on Day 21
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in static mode (PHASE A) | End of the 3-hour period on Day 28
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in dynamic mode (PHASE B) | End of the 3-hour period on Day 7
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in dynamic mode (PHASE B) | End of the 3-hour period on Day 14
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in dynamic mode (PHASE B) | End of the 3-hour period on Day 21
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under
Forward slippage in dynamic mode (PHASE B) | End of the 3-hour period on Day 28
  Measurement of forward slippage (mm) of the pelvis in relation to the backrest of the chair. This assessment will be made after each involuntary movement over the 3-hour observation period.Collection tools/methods :
  Go pro positioning: see face + torso Sensor positioning: 4 motion sensors record continuously throughout the sequence: one on the back of the chair, one on the thorax over the sternum, one on the anterior superior iliac spine and one on the top of the homolateral thigh.
  Motion sensor data are sent by e-mail ( .csv file), together with a timeline (word file) of the occurrence of abnormal movements. They are sent pseudonymized simultaneously to Mike Dongelmans (ALU REHAB AS, Norway) and MotionCatch / Denmark (which carries out the analysis on behalf of ALU REHAB AS). In order to mark the "involuntary movement" events on the video, the collaborator will have to be able to identify which chair it is, but then, for the forward-slippage data analysis, this will be done under

SECONDARY OUTCOMES:
Peak force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 7
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 14
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 21
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 28
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 7
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 14
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 21
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Peak force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 28
  Measurement of the peak force (F max ) exerted on the user's back during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 7
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 14
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 21
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in static mode (PHASE A) | After each involuntary movement over the 3-hour observation period on Day 28
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 7
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 14
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 21
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Maximum downward force in dynamic mode (PHASE B) | After each involuntary movement over the 3-hour observation period on Day 28
  Measurement of the maximum downward force (Newton) exerted on the user's seat during an involuntary movement. This assessment will be made after each involuntary movement over the 3-hour observation period.
Patient's comfort in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in static mode (PHASE A) | At the end of the 3-hour observation period on Day 14
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in static mode (PHASE A) | At the end of the 3-hour observation period on Day 21
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in static mode (PHASE A) | At the end of the 3-hour observation period on Day 28
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 7
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Patient's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Self-assessment of the comfort felt by the patient when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Caregiver's comfort in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Hetero-assessment of the comfort felt by the patient's caregiver when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Caregiver's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Hetero-assessment of the comfort felt by the patient's caregiver when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Caregiver's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Hetero-assessment of the comfort felt by the patient's caregiver when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Caregiver's comfort in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Hetero-assessment of the comfort felt by the patient's caregiver when using the chair (Visual Analog Scale between 0 and 100mm) at the end of each measurement phase.
Number of repositionings required in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Number of repositionings required during the test phase.
Number of repositionings required in static mode (PHASE A) | At the end of the 3-hour observation period on Day 14
  Number of repositionings required during the test phase.
Number of repositionings required in static mode (PHASE A) | At the end of the 3-hour observation period on Day 21
  Number of repositionings required during the test phase.
Number of repositionings required in static mode (PHASE A) | At the end of the 3-hour observation period on Day 28
  Number of repositionings required during the test phase.
Number of repositionings required in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 7
  Number of repositionings required during the test phase.
Number of repositionings required in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Number of repositionings required during the test phase.
Number of repositionings required in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Number of repositionings required during the test phase.
Number of repositionings required in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Number of repositionings required during the test phase.
Discomfort perceived by the caregiver in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in static mode (PHASE A) | At the end of the 3-hour observation period on Day 14
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in static mode (PHASE A) | At the end of the 3-hour observation period on Day 21
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in static mode (PHASE A) | At the end of the 3-hour observation period on Day 28
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 7
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Discomfort perceived by the caregiver in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Caregiver's self-assessment of the discomfort felt over the observation period using a Visual Analog Scale scale from 0 to 100mm.
Safety as perceived by the caregiver/carer in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in static mode (PHASE A) | At the end of the 3-hour observation period on Day 14
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in static mode (PHASE A) | At the end of the 3-hour observation period on Day 21
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in static mode (PHASE A) | At the end of the 3-hour observation period on Day 28
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 7
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Safety as perceived by the caregiver/carer in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Hetero-evaluation by Visual Analog Scale scale (0-100mm) of the safety felt by the caregiver/carer when using the chair during the observation phase.
Average of peak forces exerted on the wheelchair's backrest in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in static mode (PHASE A) | At the end of the 3-hour observation period on Day 14
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in static mode (PHASE A) | At the end of the 3-hour observation period on Day 21
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in static mode (PHASE A) | At the end of the 3-hour observation period on Day 28
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 7
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's backrest in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Calculation of the average of the peak forces (Fmax) exerted on the rear support of the wheelchair.
Average of peak forces exerted on the wheelchair's seat in static mode (PHASE A) | At the end of the 3-hour observation period on Day 7
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in static mode (PHASE A) | At the end of the 3-hour observation period on Day 14
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in static mode (PHASE A) | At the end of the 3-hour observation period on Day 21
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in static mode (PHASE A) | At the end of the 3-hour observation period on Day 28
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 7
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 14
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 21
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.
Average of peak forces exerted on the wheelchair's seat in dynamic mode (PHASE B) | At the end of the 3-hour observation period on Day 28
  Calculation of the average of the peak forces (Fmax) exerted on the seat of the wheelchair measured for all involuntary movements.

OTHER OUTCOMES:
Sex | Day 0
  The sex of each patient will be recorded as MALE/FEMALE/NON-BINARY
Age | Day 0
  The age of each patient will be recorded in YEARS
Height | Day 0
  The height of each patient will be recorded in centimeters
Weight | Day 0
  The weight of each patient will be recorded in kilograms
Body mass index | Day 0
  The patient's body mass index (= kg/m2 ) will be calculated via a computerized procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Anissa MEGZARI, Study Director — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France